CLINICAL TRIAL: NCT05176197
Title: Effects of Almonds on Glycemia in Adults With Elevated Hemoglobin A1c Concentrations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Purdue University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Richard Mattes, Professor, Nutrition Sciences, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 055-055
Record Dates: First submitted 2021-11-23; First posted 2022-01-04 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Glucose Intolerance; Glucose Metabolism Disorders (Including Diabetes Mellitus)
MeSH Terms: conditions — Glucose Intolerance; Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond Group (Experimental): Participants will consume almonds every day for 16 weeks, but will not be allowed to consume any other nuts or nut products.
  Interventions: Other: Almond
- Control Group (Experimental): Participants will consume pretzels every day for 16 weeks, but will not be allowed to consume any other nuts or nut products.
  Interventions: Other: Control

INTERVENTIONS:
Other: Almond — Participants will consume almonds every day for 16 weeks.
  Arms: Almond Group
Other: Control — Participants will consume pretzels every day for 16 weeks.
  Arms: Control Group

SUMMARY:
This study will examine the effects of regular almond consumption by individuals with elevated HbA1c on long-term glycemic control.

DETAILED DESCRIPTION:
Globally, it is projected that 418 million people will have impaired glucose tolerance by 2025. In the US, an estimated 34 million Americans have diabetes and 88 million, 33% of adults, have pre-diabetes. Impaired glucose tolerance is now manifesting in young adults where 20% of those 12-18 years of age have prediabetes. The current prevalence of Type 2 diabetes is over 8%, but it is projected that up to a third of Americans will develop diabetes in their lifetime. Additionally, the total annual cost of diabetes is approximately $327 which accounts for 25% of all US health care costs. Moreover, the costs rose 60% from 2007 to 2017 and this trend is continuing.

Diet is the preferred approach for management for this diet-related chronic disorder. Accumulating evidence suggests almond consumption decreases postprandial glycemia and may evoke a second meal effect, especially when they are consumed at breakfast or as an afternoon snack, which may aid in long-term glycemic control. Additionally, almond consumption can decrease total and LDL cholesterol, resulting in lower peripheral insulin resistance and cardiometabolic complications from type 2 diabetes mellitus. However, there is mixed evidence on the effects of almond consumption on HbA1c, a clinically important endpoint that provides a reliable measure of long-term glycemia and is correlated with risk of complications from diabetes. Thus, the investigators hypothesize a beneficial effect of regular almond consumption on long-term glycemic control in individuals with elevated baseline HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c >5.7%
* BMI >20 kg/M^2
* Prefer no use of medications, but if on medication, must have been on a stable dose for 3 months and plan to remain at the same level for the duration of the trial.
* Healthy, good dentition
* No nut allergies
* >4.0 eating events per day
* >=1 low nutrient density snack/d
* No allergy to chocolate

Exclusion Criteria:

* HbA1c within normal range
* BMI <20 kg/M^2
* Nut allergies
* Smoker
* Pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline
Change in HbA1c | 16 weeks
  HbA1c % change

SECONDARY OUTCOMES:
Glucose response to a meal tolerance test | Baseline and week 16
  mg/dl
Insulin response to a meal tolerance test | Baseline and week 16
  mmol/L
Chronic glycemia | Baseline, week 8 and week 16
  mg/dl
Food intake | Two days (one week day and one weekend day) at screening, week 8 and week 16.
  kcal
Body weight | Screening, baseline, week 4, week 8, week 12, and week 16
  Kilograms (kg)
Body composition | Baseline, week 16
  Percentage (%)
Hedonic survey | Baseline, week 4, week 8, week 12. week 16
  mm on a VAS

OTHER OUTCOMES:
Compliance - Vitamin E | Baseline, week 8 and week 16.
  mg/L
Compliance - fatty acid profile | Baseline, week 8 and week 16
  % fatty acid composition

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue Univeristy, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No